CLINICAL TRIAL: NCT04515927
Title: An Open-label, Single-arm Study Evaluated the Efficacy and Safety of JS002 in Patients With Homozygous Familial Hypercholesterolemia
Brief Title: To Evaluate the Efficacy and Safety of JS002 in HoFH Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS002-004
Record Dates: First submitted 2020-08-11; First posted 2020-08-17 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Hyperlipemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- subcutaneous injection of JS002, 450mg, Q4W, 3/13 times. (Experimental)
  Interventions: Drug: JS002

INTERVENTIONS:
Drug: JS002 — Biological: JS002 Administered by subcutaneous injection

SUMMARY:
JS002 is a recombinant human anti-PCSK9 monoclonal antibody. This phase II open-label, single-arm study aims to evaluate the efficacy and safety of JS002 in patients with homozygous familial hypercholesterolemia A dose group (450 mg) was set up in this study.Thirty subjects are planned to be enrolled.

Each subject required a maximum of 6 weeks of screening, 52 weeks of treatment, and 8 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Age ≥12 and ≤75 years old;
3. Weight ≥40kg at the time of screening
4. Patients diagnosed with HoFH
5. Low-density lipoprotein cholesterol (LDL-C) level ≥3.4mmol/L at the time of screening
6. Fasting triglycerides ≤4.5 mmol/L;

Exclusion Criteria:

1. History of NYHA class III-IV heart failure or EF<30%
2. History of uncontrolled arrhythmia within 3 months
3. History of MI,UA, PCI or CABG, stroke within 3 months.
4. History of DVT or pulmonary embolism within 3 months.
5. Planned cardiac surgery or revascularization.
6. Uncontrolled hypertension.
7. Uncontrolled diabetes mellitius (HbA1c>8.0%）.
8. Other conditions that the researchers considered inappropriate to participate in the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of effectiveness | JS002 is administered subcutaneously every 4 weeks, from 12 or 52 weeks after initial administration
  Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) at Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital Capital Medical University, Beijing, Beijing Municipality, China